CLINICAL TRIAL: NCT05419687
Title: Violence Against Health Care Workers: Understanding Context Through Citizen Science and Measuring a De-escalation Training Intervention Effectiveness in Eastern Democratic Republic of Congo and Iraq
Brief Title: Violence Against Health Care Workers in Fragile Settings
Acronym: VIA-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: International Committee of the Red Cross (ICRC) (Unknown); Catholic University of Bukavu, Democratic Republic of Congo (Unknown); Al-Mustansiriyah University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 70198
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-09

CONDITIONS: Workplace Violence
Keywords: de-escalating; violence prevention; behavioral symptoms; code of conduct
MeSH Terms: conditions — Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: The SW-RCTs will consist of 11 sequences (11 different possibilities of timing and sequencing the introduction of the intervention components), and a maximum of four intervention periods, combining an individual de-escalating training intervention followed by a refreshment training in the form of a collaborative learning and a code of conduct board level intervention with an overall study duration of 24 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Only the statistician and the PI will be aware of the allocation order sequence, while the country co-investigators will be blinded to the allocation sequence and only the next health facility/secondary hospital randomized for roll out will be revealed at each crossover intervention implementation time point. The outcome assessors will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Arm 1 De-escalating violence training (Experimental): The de-escalating violence training intervention will be introduced after a pre-interventional period of 3 months. A refreshment training will be introduced at month 11.
  Interventions: Behavioral: Training in de-escalating violence
- Arm 2 De-escalating violence training (Experimental): The de-escalating violence training intervention will be introduced before the second observation period at month 11. A refreshment training will be introduced at month 18.
  Interventions: Behavioral: Training in de-escalating violence
- Arm 3 De-escalating violence training (Experimental): The de-escalating violence training intervention will be introduced before the third observation period at month 18.
  Interventions: Behavioral: Training in de-escalating violence
- Arm 4 De-escalating violence training + Code of conduct (Experimental): The de-escalating violence training intervention will be introduced after a pre-interventional period of 3 months. The code of conduct via a warning board will be introduced at month 11. A refreshment training will be introduced at month 18.
  Interventions: Behavioral: Training in de-escalating violence; Behavioral: Code of conduct delivered via a warning board
- Arm 5 De-escalating violence training + Code of conduct (Experimental): The de-escalating violence training intervention and the code of conduct via a warning board will be simultaneously introduced at month 11. A refreshment training will be introduced at month 18.
  Interventions: Behavioral: Training in de-escalating violence; Behavioral: Code of conduct delivered via a warning board
- Arm 6 Code of conduct + De-escalating violence training (Experimental): The code of conduct via a warning board will be introduced at month 11. The de-escalating violence training intervention will be introduced at month 18.
  Interventions: Behavioral: Training in de-escalating violence; Behavioral: Code of conduct delivered via a warning board
- Arm 7 De-escalating violence training + Code of conduct (Experimental): The de-escalating violence training intervention is introduced after a pre-interventional period of 3 months. The code of conduct via a warning board and a refreshment training will be simultaneously introduced at month 18.
  Interventions: Behavioral: Training in de-escalating violence; Behavioral: Code of conduct delivered via a warning board
- Arm 8 De-escalating violence training + Code of conduct (Experimental): The de-escalating violence training intervention will be introduced before the second observation period at month 11. The code of conduct via a warning board and a refreshment training will be simultaneously introduced at month 18.
  Interventions: Behavioral: Training in de-escalating violence; Behavioral: Code of conduct delivered via a warning board
- Arm 9 De-escalating violence training + Code of conduct (Experimental): The code of conduct via a warning board and the violence de-escalating training will be simultaneously introduced at month 18.
  Interventions: Behavioral: Training in de-escalating violence; Behavioral: Code of conduct delivered via a warning board
- Arm 10 Code of conduct (Experimental): The code of conduct via a warning board will be introduced at month 11.
  Interventions: Behavioral: Code of conduct delivered via a warning board
- Arm 11 Code of conduct (Experimental): The code of conduct via a warning board will be introduced at month 18.
  Interventions: Behavioral: Code of conduct delivered via a warning board

INTERVENTIONS:
Behavioral: Training in de-escalating violence — * Individual educational component through a de-escalating violence training for health care workers (verbal and non-verbal de-escalating techniques)
  * Refreshment training in the form of collaborative learning
  Arms: Arm 1 De-escalating violence training; Arm 2 De-escalating violence training; Arm 3 De-escalating violence training; Arm 4 De-escalating violence training + Code of conduct; Arm 5 De-escalating violence training + Code of conduct; Arm 6 Code of conduct + De-escalating violence training; Arm 7 De-escalating violence training + Code of conduct; Arm 8 De-escalating violence training + Code of conduct; Arm 9 De-escalating violence training + Code of conduct
Behavioral: Code of conduct delivered via a warning board — A publicly displayed code of conduct (a co-designed set of rules) for both HCWs and clients, delivered via a warning board at the level of the health facilities and secondary hospitals
  Arms: Arm 10 Code of conduct; Arm 11 Code of conduct; Arm 4 De-escalating violence training + Code of conduct; Arm 5 De-escalating violence training + Code of conduct; Arm 6 Code of conduct + De-escalating violence training; Arm 7 De-escalating violence training + Code of conduct; Arm 8 De-escalating violence training + Code of conduct; Arm 9 De-escalating violence training + Code of conduct

SUMMARY:
The general objective of the project is to assess whether a violence de-escalating training for health professionals and of a publicly displayed Code of Conduct (a set of rules developed through a citizen science and co-design approach) for both health professionals and clients at the level of the health facility, can reduce the incidence and severity of episodes of violence, and to identify the most cost-effective way to implement these interventions in rural Democratic Republic of Congo (DRC) and in the mega city of Baghdad, Iraq.

DETAILED DESCRIPTION:
The study will adopt a stepped-wedge cluster-randomized intervention trial (SW-CRT) design to assess the two intervention components, a violence de-escalating training and the implementation of the code of conduct co-developed during the formative qualitative phase. The study will adopt a closed cohort with repeated measurements on the same participants (nurses in DRC and junior doctors in Baghdad) and will involve the unidirectional transition of each enrolled cluster (health facilities in DRC and secondary hospitals in Baghdad) from the control (no intervention) to the intervention sequence in a randomized sequential manner according to a predefined roll out process.

ELIGIBILITY:
Inclusion Criteria:

* HCWs from selected participating health facilities in DRC, junior doctors during their first year resident and permanent health care staff from participating secondary hospitals in Iraq
* HCWs and junior medical doctors and permanent health care staff must have been employed/ or worked as HCW/ medical doctors or as permanent health care staff for at least 6 months
* All above participants must have completed the written informed consent

Exclusion Criteria:

* Age <18 years; cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 798 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of self-reported non-physical aggression | 6 months
  Number of self-reported non-physical aggression (verbal abuse, threats, ironic language, provocative or aggressive body language etc.) during the fulfillment of a professional activity in the last 6 months
Incidence and severity of self-reported physical aggression | 6 months
  Number of self-reported physical aggression during the fulfillment of a professional activity in the last 6 months

SECONDARY OUTCOMES:
Level of confidence in coping with patient aggression | 0, 6, 12, 18 months
  Instrument "Clinicians confidence in coping with patient aggression (CCPAI) (Thackreys, 1987)"
Level of post-traumatic stress disorders (PTSD) among HCWs | 0, 6, 12, 18 months
  Instrument "Post-traumatic stress disorder PTSD Checklist for DSM-5 (PCL-5)) (Weathers, F.W. et al. 2013)"
Level of burnout among HCWs | 0, 6, 12, 18 months
  Instrument "Level of burnout" (Malach 2005), burnout measure short version (BMS). The ten-item version of the BMS are evaluated on 7-point frequency scales, with a score of 4 or above indicating burnout.
Psychological empathy among HCWs | 0, 6, 12, 18 months
  Instrument "Jefferson scale of physician empathy (Hojat M et al. 2007)"
Absenteeism | 0, 6, 12, 18 months
  Number of sick leave spells taken by the HCWs during the study period
Intent to leave among HCWs | 0, 6, 12, 18 months
  The shortened, six-item version of the turnover intention scale (TIS-6) (Bothma & Roodt 2013), will be used to assess turnover intentions and as well as to predict actual turnover among HCWs. The TIS-6 scale is scored on a five-point Likert-type scale with scores ranging from 1 (never) to 5 ( always). A high score indicates stronger turnover intention.
Economic cost of the intervention | 18 months
  Two types of costs will be considered: 1) direct costs of the intervention (e.g training costs, space or rent costs, costs to develop the code of conduct) and 2) direct costs due to health system disruption (e.g. health care services foregone or postponed, material etc.), cost incurred by the HCWs as a consequence of violent episodes including direct medical costs (e.g. hospital stay cost, consultation costs, laboratory costs), non-medical costs (e.g. transportation, meals etc.), and indirect costs (e.g. absenteeism, presenteeism).
Productivity loss (presenteeism) | 18 months
  Work Limitation questionnaire (WLQ) (Lerner D. et al. 2002). The WLQ consists of eight items investigating four domains (time management, physical tasks, mental-interpersonal tasks, and output tasks), which are calculated into scores ranging from 0 (no limitations) to 100 (highest limitations).
Health care workers health-related quality of life | 0, 6, 12, 18 months
  European Quality of Life-5 Dimensions (EuroQol EQ-5D-5L) (Devlin NJ et al. 2017). The EQ-5D-5L questionnaire is self-assessed and it measures health outcomes on five dimensions (mobility, self-care, daily activities, pain/discomfort, and depression/anxiety) with five levels ranging from none to major complaints. Scores range from 0 (death) to 1 (full health).

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Merten, MD MPH PhD, Principal Investigator — Swiss Tropical and Public Health Institute (Swiss TPH)
Locations (2):
- Catholic University of Bukavu, School of Public Health, Bukavu, Democratic Republic of the Congo
- Al-Mustansiriya University, Baghdad, Iraq

REFERENCES:
- [Background] Elrha, International Committee of the Red Cross (ICRC), RAND Europe. Researching Violence Against Health Care: Gaps and Priorities. 2020
- [Background] Leach, Brandi, Emily Ryen Gloinson, Alex Sutherland, and Michael Whitmore, Reviewing the Evidence Base for De-escalation Training: A Rapid Evidence Assessment. Santa Monica, CA: RAND Corporation, 2019.
- [Background] Geoffrion S, Hills DJ, Ross HM, Pich J, Hill AT, Dalsbo TK, Riahi S, Martinez-Jarreta B, Guay S. Education and training for preventing and minimizing workplace aggression directed toward healthcare workers. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD011860. doi: 10.1002/14651858.CD011860.pub2. PMID 32898304
- [Derived] Ferrari G, Lwamushi SM, Balaluka GB, Lafta RK, Schindler C, Bugugu D, Lurhangire E, Tediosi F, Mendoza JR, Merten S. Understanding context of violence against healthcare through citizen science and evaluating the effectiveness of a co-designed code of conduct and of a tailored de-escalation of violence training in Eastern Democratic Republic of Congo and Iraq: a study protocol for a stepped wedge randomized controlled trial. Trials. 2023 Dec 19;24(1):814. doi: 10.1186/s13063-023-07839-3. PMID 38110997